CLINICAL TRIAL: NCT00178438
Title: A Prospective Trial of Wireless Capsule Endoscopy in Small-Bowel Crohn's Disease
Brief Title: Wireless Capsule Endoscopy in Small-Bowel Crohn's Disease
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RSRB # 10455
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Crohn's Disease
Keywords: capsule endoscopy in small bowel
MeSH Terms: conditions — Crohn Disease | interventions — Capsule Endoscopy

INTERVENTIONS:
Device: Capsule Endoscopy

SUMMARY:
The purpose of this study is to determine the best role for capsule endoscopy in diagnosing Crohn's disease.

DETAILED DESCRIPTION:
Wireless capsule endoscopy (CE) is a Food and Drug Administration (FDA) approved technology that allows viewing of the entire small-bowel. Capsule endoscopy involves swallowing a pill-sized camera that sends images to a data recorder worn on a vest. Because Crohn's disease (CD) often involves the small bowel, we would like to find out if capsule endoscopy is useful in diagnosing small-bowel Crohn's disease. Current methods for diagnosing small-bowel Crohn's disease include colonoscopy, esophagogastroduodenoscopy (EGD), enteroscopy (ENT), single contrast barium small-bowel follow through (SBFT), and double contrast small-bowel enteroclysis (SBE), but these tests are unable to identify the presence or extent of small-bowel disease in many patients.

ELIGIBILITY:
Inclusion Criteria:

* English speaking adult patients (>18 years old) with known Crohn's disease

Exclusion Criteria:

* Severe medical or psychiatric co-morbidities
* Active swallowing problems
* Bowel obstruction
* History of stricture or fistula
* Pregnancy
* Taking aspirin/non-steroidal anti-inflammatory drug (NSAID) or potassium chloride (KCl) within 4 weeks prior to the colonoscopy and anytime after colonoscopy
* Inability to consent
* Exclusion of patients whose colonoscopy was done for reasons other than signs/symptoms suggestive of Crohn's disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-06; Study Completion 2006-06

PRIMARY OUTCOMES:
Compare capsule endoscopy (CE) finding with traditional findings (colonoscopy and small-bowel follow through [SBFT]) in patients with known Crohn's disease

SECONDARY OUTCOMES:
Evaluate the extent and severity of CE determined small-bowel involvement in patients with known Crohn's disease

CONTACTS AND LOCATIONS:
Overall Officials: Parvez S Mantry, MD, Principal Investigator — University of Rochester Medical Center, Digestive and Liver Disease Unit
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States